CLINICAL TRIAL: NCT05709652
Title: Impact of Fast Gantry Rotation Cardiac CT Angiography on Coronary Motion Artifacts in the Absence of β-Blocker Premedication in Patients Undergoing Aortic Stenosis Workup: a Single-centre Randomized Controlled Trial
Brief Title: Impact of Fast-rotation Coronary CT in Patients Undergoing Aortic Stenosis Workup
Acronym: FAST-CCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David C. Rotzinger (Other)
Responsible Party: Sponsor-Investigator, David C. Rotzinger, MD, PhD, head of cardiovascular and thoracic radiology, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BPR526
Record Dates: First submitted 2023-01-11; First posted 2023-02-02 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Coronary Stenosis; Aortic Valve Stenosis; Cardiovascular Diseases
Keywords: Computed Tomography Angiography; Artifacts; Diagnostic imaging; Image Processing, Computer-Assisted
MeSH Terms: conditions — Coronary Stenosis; Aortic Valve Stenosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients subjected to aortic CTA with a gantry revolution time of 0.23 sec
  Interventions: Diagnostic Test: Aortic CTA, .23s
- Control (Active Comparator): Patients subjected to aortic CTA with a gantry revolution time of 0.28 sec
  Interventions: Diagnostic Test: Aortic CTA, .28s

INTERVENTIONS:
Diagnostic Test: Aortic CTA, .23s — Aortic CTA performed with short (0.23 sec) gantry rotation time.
  Other Names: GE Healthcare, Revolution Apex, cardiac and aortic CT angiography with 230 ms rotation time
  Arms: Experimental
Diagnostic Test: Aortic CTA, .28s — Aortic CTA performed with standard (.28 sec) gantry rotation time.
  Other Names: GE Healthcare, Revolution Apex, cardiac and aortic CT angiography with 280 ms rotation time
  Arms: Control

SUMMARY:
This study aims to evaluate the clinical value of a novel CT gantry supporting a .23 second rotation time and systematically compare it with 0.23 second rotation time, in patients with clinically indicated aortic CTA in the workup of aortic stenosis. Patients will be randomly assigned .23 or .28 sec rotation time CTA. Coronary artery interpretability rates will be determined in both groups.

DETAILED DESCRIPTION:
Coronary artery analysis is an essential component of cardiac CT, but is often challenging without beta-blocker use. CT's technological advances are continuously evolving, paving the way for safer and more accurate diagnoses. Part of these innovations is the development of faster rotation speeds (0.23 sec/rotation), which is expected to allow for heart rate-independent CCTA.

Patients subjected to aortic stenosis workup routinely undergo invasive coronary angiography (ICA) in the catheterization laboratory, voiding the need to control the heart rate at the time of cardiac CT because aortic valve measurements can be performed even at higher heart rate. Still, cardiac CT in this context is performed with ECG-gating, and attempting to evaluate coronary arteries is possible without interfering with clinical decisions. Also, the existing literature advocates the use of gantry rotation speeds of at least 0.5 sec/rotation; consequently, the use of 0.28 versus 0.23 sec/rotation for this study will comply with current guidelines and will have no detrimental impact on patient management. This study aims to evaluate coronary artery interpretability in patients subjected to cardiac CT for the anatomical assessment of aortic valve stenosis prior to endovascular (transcatheter aortic valve implantation [TAVI]) or surgical therapy.

Patients will be enrolled after providing written, informed consent, and will be randomly assigned either to the test (0.23 sec rotation time) or control group (0.28 sec rotation).

The participants concerned are not subjected to any additional invasive or stressful procedure compared with those undergoing aortic stenosis workup in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Subjected to cardiac CT due to known or suspected aortic valve stenosis

Exclusion Criteria:

* Patients unable to hold their breath, deaf or visually impaired
* Estimated glomerular filtration rate (eGFR) of <30 mL/min
* Hemodynamic instability or cardiogenic shock, Acute pulmonary edema, Exacerbated chronic obstructive pulmonary disease, Pregnant and breast-feeding women
* Patients with prior coronary artery bypass grafting (CABG)
* Patient incapable of discernment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Interpretable CTA rate per patient | Up to 90 days
  Number of patients with diagnostic image quality for coronary artery disease

SECONDARY OUTCOMES:
Interpretable CTA rate, per segment | Up to 90 days
  Number of segments with diagnostic image quality for coronary artery disease
CTA performance to measure diameter stenosis, using invasive coronary angiography as gold standard | Coronary angiography performed withing 30 days of CTA
  CTA's diagnostic accuracy for coronary occlusive disease
Relationship between heart rate and non-diagnostic CTA | Up to 90 days
  Correlation between of heart rate (in BPM) and the presence of any uninterpretable coronary segment on CTA
Quantitative image quality (contrast to noise ratio) | Up to 90 days
  Comparison of contrast to noise ratio between both groups
Radiation dose per patient | Up to 90 days
  Effective dose (mSv) comparison between both groups

CONTACTS AND LOCATIONS:
Overall Officials: David C. Rotzinger, MD, PhD, Principal Investigator — CHUV
Locations (1):
- Lausanne University Hospital (CHUV), Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fahrni G, Gullo G, Touray A, Fournier S, Jouannic AM, Lu H, Racine D, Muller O, Pozzessere C, Qanadli SD, Rotzinger DC. Investigating the Influence of High-Speed Gantry Rotation in Cardiac CT on Motion Artifacts in Aortic Stenosis Patients Not Premedicated with beta-Blockers: The FAST-CCT Randomized Trial Protocol. J Cardiovasc Dev Dis. 2023 Oct 12;10(10):424. doi: 10.3390/jcdd10100424. PMID 37887871